CLINICAL TRIAL: NCT06228911
Title: Increased Blood Glucose Levels After Steroid Injection Into Osteoarthritic Knee in Diabetic Patients' Type 2
Brief Title: Increased Blood Glucose Levels After Steroid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Diaa Haj Ali, Medical Doctor Diaa Haj Ali, Syrian Private University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: GH; 5615
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee; Diabete Type 2
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus, Type 2 | interventions — Steroids; Triamcinolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insulin treated group (Experimental)
  Interventions: Drug: steroid (triamcinolone)
- non-insulin treated groups (Experimental)
  Interventions: Drug: steroid (triamcinolone)

INTERVENTIONS:
Drug: steroid (triamcinolone) — triamcinolone is a synthetic corticosteroid medication used topically to treat various skin conditions, to relieve the discomfort of mouth sores, and by injection into joints to treat various joint conditions

SUMMARY:
a sample of 600 patients diagnosed as Knee osteoarthritis injected with 40 mg triamcinolone, recorded their morning fasting blood glucose levels for 7 days before injection used as the baseline blood glucose level, which was compared with FBS levels for 14 days after steroid injection. Our study compared the differences in blood glucose changes between HbA1c >7% and HbA1c ≤7% groups and those between insulin and non-insulin treated groups.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years, patients with knee osteoarthritis diagnosed according to American College of Rheumatology (ACR) Criteria (17), and grade1-3 in Kallgren-Laurence radiographic scale (18), whom failed to response to medical treatment including paracetamol and nonsteroidal anti-inflammatory medication, and to physical therapy, checking their blood glucose values daily.

Exclusion Criteria:

Patients who were unable to provide consent, patients had any contraindications to corticosteroids, patients who had received oral corticosteroid in the past 6 months or corticosteroid injection in the previous 3 months, patients who had no monitoring HbA1c level before injection or also whom had not monitor blood glucose levels before or after injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
high blood glucose | 3 years
  glucose increases after steroid dose
low blood glucose | 3 years
  glucose decreases after steroid dose

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Damascus University, Syria, Damascus, Syria